CLINICAL TRIAL: NCT04718350
Title: Comparison of Intravenous Levosimendan and Inhalational Milrinone in High Risk Cardiac Patients With Pulmonary Hypertension
Brief Title: Treatment of Pulmonary Hypertension in High-risk Cardiac Surgery Patients Using Inhalational and Intravenous Agents
Acronym: levos-milr
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Professor of Anesthesiology, Aretaieion University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: levo-milri
Record Dates: First submitted 2021-01-16; First posted 2021-01-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Hypertension, Pulmonary; Cardiac Failure; Pulmonary Vascular Resistance Abnormality
Keywords: pulmonary vascular resistance; pulmonary hypertension; vasodilators; milrinone; levosimendan; cardiopulmonary bypass
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous administration of Levosimendan at a dosage of 6 mcg/kg after induction of anesthesia (Active Comparator): in this group, 6 mcg/kg of levosimendan will be administered intravenously after anesthesia induction, aiming at prevention of pulmonary hypertension post bypass
  Interventions: Drug: levosimendan at a dose of 6 mcg/kg
- Inhalational administration of Milrinone at a dosage of 50 mcg/kg after induction of anesthesia (Active Comparator): in this group, 50 mcg/kg of milrinone will be administered via inhalation after anesthesia induction, aiming at prevention of pulmonary hypertension post bypass
  Interventions: Drug: milrinone at a dose of 50 mcg/kg

INTERVENTIONS:
Drug: levosimendan at a dose of 6 mcg/kg — levosimendan will be administered intravenously at a dose of 6 mcg/kg after anesthesia induction
  Other Names: Group Levo
  Arms: Intravenous administration of Levosimendan at a dosage of 6 mcg/kg after induction of anesthesia
Drug: milrinone at a dose of 50 mcg/kg — milrinone will be administered via inhalation at a dose of 50 mcg/kg after anesthesia induction
  Other Names: Group Milri
  Arms: Inhalational administration of Milrinone at a dosage of 50 mcg/kg after induction of anesthesia

SUMMARY:
The aim of this study is to examine and compare the effect of Levosimendan and Milrinone administered intravenously and via inhalation respectively in cardiac surgery patients with pulmonary hypertension and right ventricular dysfunction.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is a pathophysiological disorder hemodynamically characterized by increased pulmonary vascular resistance and pressure. This can lead to right ventricle pressure overload and failure, which is worsened by cardiopulmonary bypass (CPB) and extracorporeal circulation and is accompanied by high rates of morbidity and mortality in cardiac surgery patients. Pharmacological agents used to decrease pulmonary vascular resistance and right ventricle afterload are prostaglandins, iloprost, milrinone, nitric oxide (NO) and recently Levosimendan. These agents can be administered intravenously or via inhalation.

In this study, the intravenous administration of Levosimendan will be compared with the inhalational use of milrinone in patients with pulmonary hypertension undergoing cardiac surgery.

In this setting, 40 patients with PH caused by left sided heart disease, will be assigned into two groups:

GROUP A: Intravenous administration of Levosimendan in dosage 6mcg/kg after induction of anesthesia.

GROUP B: Inhalational administration of milrinone in dosage 50mcg/kg after induction of anesthesia.

Before and after the administration of the drug, heart function will be evaluated by hemodynamic measurements obtained by the Swan-Ganz catheter. These parameters will be heart rate (HR), blood pressure (BP), mean pulmonary arterial pressure (MPAP), central venous pressure (CVP), cardiac output (CO), pulmonary capillary wedge pressure (PCWP), cardiac index (CI), systemic vascular resistance (SVR), pulmonary vascular resistance (PVR). Transthoracic echocardiography (TTE) and transoesophageal echocardiography (TOE) will also be used.

This study will lead to conclusions regarding the effectiveness of intravenous administration of Levosimendan and inhalational use of Milrinone in the treatment of right heart failure and PH in cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with pulmonary hypertension due to left ventricular dysfunction based on echocardiographic diagnosis preoperatively
* elective cardiac surgery

Exclusion Criteria:

* primary pulmonary hypertension
* thromboembolic disease
* chronic obstructive pulmonary disease
* emergency surgery
* redo surgery
* inability to consent to the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
change from baseline in mean pulmonary arterial pressure (MPAP) | 20 minutes after vasodilator administration, at the end of surgery and 2 hours after Intensive Care Unit (ICU) admission
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in pulmonary vascular resistance (PVR) | 20 minutes after vasodilator administration, at the end of surgery and 2 hours after Intensive Care Unit (ICU) admission
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in mean arterial pressure (MAP) | 20 minutes after vasodilator administration, at the end of surgery and 2 hours after Intensive Care Unit (ICU) admission
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in systemic vascular resistance (SVR) | 20 minutes after vasodilator administration, at the end of surgery and 2 hours after Intensive Care Unit (ICU) admission
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in pulmonary capillary wedge pressure (PCWP) | 20 minutes after vasodilator administration, at the end of surgery and 2 hours after Intensive Care Unit (ICU) admission
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in cardiac output (CO) | 20 minutes after vasodilator administration, at the end of surgery and 2 hours after Intensive Care Unit (ICU) admission
  a Swan-Ganz catheter will be used for hemodynamic measurements
change from baseline in tricuspid annular plane systolic excursion (TAPSE) | 20 minutes after vasodilator administration, at the end of surgery and 2 hours after Intensive Care Unit (ICU) admission
  transthoracic and transesophageal echocardiography will be used for echocardiographic measurements
change from baseline in fractional area change | 20 minutes after vasodilator administration, at the end of surgery and 2 hours after Intensive Care Unit (ICU) admission
  transthoracic and transesophageal echocardiography will be used for echocardiographic measurements
length of ICU stay | postoperatively, an average period of 7-10 days
  duration of patient stay in ICU in days
hospitalization time | postoperatively, up to 20 days after the operation
  duration of hospital stay after surgery in days

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, DESA, Principal Investigator — Aretaieion University Hospital
Locations (1):
- Onassis Cardiac Surgery Center, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Theodoraki K, Thanopoulos A, Rellia P, Leontiadis E, Zarkalis D, Perreas K, Antoniou T. A retrospective comparison of inhaled milrinone and iloprost in post-bypass pulmonary hypertension. Heart Vessels. 2017 Dec;32(12):1488-1497. doi: 10.1007/s00380-017-1023-2. Epub 2017 Jul 17. PMID 28717881
- [Background] Haddad F, Couture P, Tousignant C, Denault AY. The right ventricle in cardiac surgery, a perioperative perspective: II. Pathophysiology, clinical importance, and management. Anesth Analg. 2009 Feb;108(2):422-33. doi: 10.1213/ane.0b013e31818d8b92. PMID 19151265
- [Background] Hansen MS, Andersen A, Nielsen-Kudsk JE. Levosimendan in pulmonary hypertension and right heart failure. Pulm Circ. 2018 Jul-Sep;8(3):2045894018790905. doi: 10.1177/2045894018790905. Epub 2018 Jul 6. PMID 29979110
- [Background] Kundra TS, Nagaraja PS, Bharathi KS, Kaur P, Manjunatha N. Inhaled levosimendan versus intravenous levosimendan in patients with pulmonary hypertension undergoing mitral valve replacement. Ann Card Anaesth. 2018 Jul-Sep;21(3):328-332. doi: 10.4103/aca.ACA_19_18. PMID 30052230
- [Background] Elhassan A, Essandoh M. Inhaled Levosimendan for Pulmonary Hypertension Treatment During Cardiac Surgery: A Novel Application to Avoid Systemic Hypotension. J Cardiothorac Vasc Anesth. 2019 Apr;33(4):1169-1170. doi: 10.1053/j.jvca.2018.11.039. Epub 2018 Nov 28. No abstract available. PMID 30612930